CLINICAL TRIAL: NCT07029802
Title: Development of a Novel Evaluation Scale of Mental Body Representation (MBR) for Adults With Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PMR-2023-32512
Record Dates: First submitted 2025-05-30; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with SCI
  Interventions: Other: No intervention
- Uninjured participants
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
The purpose of this study is twofold: (1) Develop a new evaluation scale for mental body representations (MBR, i.e., body awareness and visuospatial body maps) for adults with spinal cord injury (SCI) with and without neuropathic pain. (2) Assess the psychometric properties of usability, reliability, and validity of the new evaluation scale This is a cross-sectional observational study design. For Aim 1, this study will involve initial item generation for a novel MBR evaluation scale for SCI through email communication, and individual interviews proctored remotely through Zoom, or, if preferred by the participant, in-person. For Aim 2, the study will include a Zoom call for consenting and questionnaires, as well as an in-person visit where participants will be tested with the new SCI-BodyMap evaluation scale, and a questionnaire asking about the usability and satisfaction of the new evaluation scale.

ELIGIBILITY:
Inclusion Criteria:

Control group

* Uninjured adults (from the contact list with the Brain Body Mind lab or through fliers or StudyFinder)
* 18+ years old adults

SCI group

* 18+ years old, participants with an incomplete or complete SCI of ≥ 1 year
* medically stable
* able to read and understand English
* having access to the internet/iPad/computer/phone and willing to come in for an in-person testing at the University of Minnesota.

Exclusion Criteria:

SCI group

* Uncontrolled seizure disorder;
* cognitive impairment and/or communicative disability (e.g., due to brain injury) preventing them from following directions or from learning;
* ventilator dependency;
* major medical complications;
* pressure ulcers hindering prolonged sitting or lying down.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For all adults with SCI in this study: 18+ years old, participants with an incomplete or complete SCI of ≥ 1 year, medically stable, able to read and understand English, having access to the internet/iPad/computer/phone and willing to come in for an in-person testing at the University of Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Reliability of the scale | 1 week
  Inter-rater reliability of the new SCI-BodyMap scale (scores from two physical or occupational therapists testing the same participants) will be evaluated with Kappa and ICC.
Validity of the scale | 1 week
  Convergent validity of the newly developed SCI-BodyMap scale for SCI will be tested with Spearman rho correlations between the new MBR scale and the Revised Body awareness scale, Multidimensional Assessment lnteroceptive Awareness-2 (MAIA- 2), lowest, average and highest neuropathic pain levels with the Numeric Pain Rating Scale (NPRS), and the NINOS-COE SCI Functional lndex/Assistive Technology Scale (SCI/Fl-AT).
establish the minimal detectable difference (MDD) | 1 week
  The Minimal Detectable Difference (MOD) will be calculated using the standard error of measurement.

SECONDARY OUTCOMES:
QQ-10 scale, to assess the usability of the new MBR scale. | 1 week
  This will be complemented by open-ended questions about the scale from the point of view of the participant with SCI and the therapists who evaluated the participant with the new scale.
SCI-related symptoms (Penn Spasm Frequency Scale | 1 week
  We will assess the frequency and severity of spasms (Penn Spasm Frequency Scale),
SCI-related symptoms (BARQ-R) | 1 week
  We will assess body awareness related to the participant's perception of tension in the body (BARQ-R)
SCI-related symptoms (MAIA-2) | 1 week
  We will assess interoceptive awareness (MAIA-2).
Physical functioning. | 1 week
  We will measure function related to basic mobility, self-care, fine motor function, and ambulation (NINOS-COE SCI/Fl-AT)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van de Winckel, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States